CLINICAL TRIAL: NCT04483024
Title: A Randomized, Double-blind, Four-arm Pilot Study to Evaluate the Effects of BRAND'S Chicken Extract and Collagen on Joint, Bone and Muscle Functions
Brief Title: Effects of Chicken Extract and Collagen on Mobility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shan May Yong (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Shan May Yong, Manager, Cerebos Pacific Limited
Organization: Cerebos Pacific Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BEC-CH-001
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Knee Osteoarthritis; Muscle Loss
MeSH Terms: conditions — Osteoarthritis, Knee; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Four-arm Pilot Study to Evaluate the Effects of Brands Chicken Extract and Collagen on Joint, Bone, and Muscle Functions
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Collagen hydrolysate and chicken extract
- Glucosamine (Active Comparator): Glucosamine hydrochloride
  Interventions: Dietary Supplement: Collagen hydrolysate and chicken extract
- Collagen hydrolysate (Experimental): 2g of hydrolyzed collagen II
  Interventions: Dietary Supplement: Collagen hydrolysate and chicken extract
- Collagen hydrolysate + chicken extract (Experimental): 2g of hydrolyzed collagen II with chicken extract
  Interventions: Dietary Supplement: Collagen hydrolysate and chicken extract

INTERVENTIONS:
Dietary Supplement: Collagen hydrolysate and chicken extract — One bottle (68mL) of collagen hydrolysate (2g) in chicken extract taken daily in the morning after meal for 24 weeks
  Other Names: BRAND'S chicken extract

SUMMARY:
A randomized, double-blind placebo-controlled trial to study the effects of chicken extract and collagen on join, bone and muscle functions in comparison to an active comparator glucosamine

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee, which entails the destruction of knee cartilage and remodeling of the adjacent bone, is one of the leading causes of disability among elderly adults. Consequences of severe knee OA, including loss of mobility and limited daily activities, affect individuals and society economically. The World Health Organization (WHO) Global Burden of Disease Study, conducted in 21 epidemiological regions worldwide, reported a 26.6% increase in the burden of knee OA from 1990 to 2010.

Current therapies for OA include various over the counter analgesics, a number of non-steroidal anti-inflammatory drugs (NSAIDs), intra-articular injections of corticosteroids or hyaluronic acid, plus tramadol and other opioid analgesics to relieve severe pain. , While these therapies can alleviate symptoms in the near term, their ultimate impact on the pathophysiologic progression of OA is limited. In addition, there are considerable side effects associated with the use of these drugs. Total joint replacement is typically the final and only effective solution for relieving pain and disability.

As a result, OA sufferers always turn to natural nutraceuticals to ease their pain and discomfort. These products are commonly used because they are well tolerated and considered safe. Nutraceuticals are defined as functional foods, natural products, or parts of food that provide medicinal, therapeutic, or health benefits, including the prevention or treatment of disease. Currently, glucosamine and chondroitin are the two most commonly used nutraceuticals in humans to alleviate pain associated with arthritis. However, recent randomized controlled trials and meta-analysis of these supplements have shown only small-to-moderate symptomatic efficacy in OA.

It therefore seems appropriate to explore other natural supplements/ingredients. There is growing interest in hydrolyzed collagen (or collagen hydrolysate [CH]) as a nutraceutical supplement because collagen-derived peptides harbor a variety of interesting biological properties. CH has been found to down-regulate inflammatory markers involved in joint inflammation and cartilage degradation such as interleukins (ILs), IL-6, IL-7, IL-9 and IL-12 as well as monocyte-chemoattractant-1 (MCP-1) in chondrocytes induced with IL-1 beta. In addition, CH reduces bone resorption in an in vitro model for regulation of osteoclastic differentiation and bone resorption by RANKL system (unpublished data).

CH has received considerable attention in relieving OA-associated symptoms. The hypothesis of how CH may reduce OA-associated symptoms includes providing bioavailable substrate (building blocks) for the collagen fibrillar network, which provides tensile strength for the matrix of articular cartilage. Oesser et al. in a series of preclinical studies, demonstrated that CH passes across the mucosal barrier in the small bowel as a complete peptide that is no longer subject to enzymatic cleavage, accumulates in cartilage tissue, and stimulates production of type II collagen (the major protein in articular cartilage) and proteoglycans in the extracellular matrix of cartilage. , , In addition to these preclinical studies, open label, comparative, and prospective, randomized, placebo-controlled clinical trials and experimental findings have been published, with several studies providing evidence of a beneficial effect on measurements of joint health from the administration of collagen hydrolysate in a variety of patient populations, mostly OA patients. , , , , , CH per day for 3 months produced an improvement in joint health or function, such as reduction in pain,11,12,14 decreased dependency on pain medications,14 and improvement in leg strength.16 Given these observations, the investigators develop a supplementation of chicken essence with additive of CH-Brands Essence of Chicken plus CH (BEC-CH). The CH is derived from chicken cartilage. It is a soluble naturally occurring matrix of hydrolyzed collagen type II, chondroitin sulfate, and hyaluronic acid. The composition is similar to that of the human articular cartilage lining found in the synovial joints. Regarding BEC, it has been consumed for decades as a health tonic for energy boosting and fatigue recovery. In fact, BEC supplementation has been clinically proven to accelerate the recovery from exercise by increasing the rate of clearance of plasma lactate and ammonia and hence reduces muscle fatigue. However, all of these data are based on supplementation of either BEC of CH per se in clinical or in in vitro settings. Thus, it is crucial to investigate the efficacy of both BEC and CH when taken in combination on joint, bone, and muscle function. To answer these questions and to investigate its tolerability and efficacy, this randomized, double-blind, four-arm pilot study is thus carried out. It is hypothesized that supplementation with BEC-CH might relieve joint discomfort, restore joint function, and also be beneficial to bone and muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female at 45 - 75 years of age
2. Subject has a body mass index range of 18.0 to 30.0 kg/m2, inclusive, and weighs at least 40 kg at screening
3. Subject agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the study.
4. Experience knee pain ≥ 3 months
5. WOMAC total pain score ≥ 6 evaluated by walking on a flat surface, descending and/or ascending stairs
6. Subject has mild-to-moderate knee osteoarthritis (OA) at grade 1 - 3 per Kellgren-Lawrence grading system
7. Experience loss in muscular strength or physical performance greater than 1 year
8. Be willing to refrain from hormone therapy and dietary supplements such as calcium, vitamin D, supplements enriched with proteins, omega-3, omega-6, glucosamine, or chondroitin during the entire study

Exclusion Criteria:

1. Inability to participate in the evaluation of the study
2. Active viral infection or bacterial infection based on clinical observations
3. Subjects with history of rheumatoid arthritis or any other inflammatory arthritis
4. Chronic medical conditions including renal dysfunctions, psychiatric disorders, or diabetes (or HbA1c > 6.5%)
5. History of stroke or myocardial infarction, mental retardation, or schizophrenia
6. Gout
7. Paget disease of bone or spinal disc herniation
8. Subjects intolerant or allergic to protein-based food or supplement
9. Anti-osteoporotic therapy in the past year
10. Intra-articular injection during previous 3 months (6 months for hyaluronic acid) applied at target knee joint (most painful knee joint at Screening visit)
11. Current corticosteroid therapy
12. Those expecting knee arthroscopy or arthroplasty
13. Life-threatening pathology (such as cancer) in remission for less than 1 year or still ongoing
14. Psychological or linguistic incapability to sign the informed consent
15. History of allergy to chicken meat
16. Pregnant or lactating women
17. Suspected or known alcohol abuse or addiction (consume ≥ 14 drinks of alcohol per week; 1 drink: ~355-mL beer or 150-mL wine)
18. Subjects with any other conditions or diseases that investigator considers not appropriate to be entered in the study
19. Subjects with active pathology that could confound interpretation of knee pain or any conditions that interfere with adherence

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC scores from baseline | 6 months
  knee joint pain
Change in Visual Analgoue Scale (VAS) pain scores from baseline | 14 days
  knee joint pain

SECONDARY OUTCOMES:
Change in Bone mass from baseline | 6 months
  Lumbar spine, left and right hip
Change in Handgrip strength from baseline | 6 months
  Average of both hands

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Nung Shih, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen CC, Chang SS, Chang CH, Hu CC, Nakao Y, Yong SM, Mandy YLO, Lim CJ, Shim EK, Shih HN. Randomized, double-blind, four-arm pilot study on the effects of chicken essence and type II collagen hydrolysate on joint, bone, and muscle functions. Nutr J. 2023 Mar 15;22(1):17. doi: 10.1186/s12937-023-00837-w. PMID 36918892